CLINICAL TRIAL: NCT04550351
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Trial to Evaluate the Safety and Tolerability of Recombinant New Coronavirus Vaccines (CHO Cells) in Healthy People Aged 60 Years and Above
Brief Title: Recombinant New Coronavirus Vaccine (CHO Cells) to Prevent SARS-CoV-2 Phase I Clinical Trial (≥60 Years Old)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LKM-2020-NCV03
Record Dates: First submitted 2020-08-16; First posted 2020-09-16 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus
Keywords: Recombinant Novel Coronavirus Vaccine
MeSH Terms: conditions — Coronavirus Infections | interventions — Biological Products; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Population I (Experimental): Population I has 20 subjects and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population I is intramuscular injection of deltoid muscle of upper arm with low dose of vaccine.
  Interventions: Biological: Biological/Vaccine: Recombinant new coronavirus vaccine (CHO cell) low-dose group
- Population II (Experimental): Population II has 20 subjects and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population II is a high-dose vaccine intramuscular injection of deltoid muscle of the upper arm.
  Interventions: Biological: Biological/Vaccine: Recombinant new coronavirus vaccine (CHO cells) high-dose group
- Population Ⅲ (Placebo Comparator): Population Ⅲ has 10 subjects and is considered negative for SARS-COV-2 and fluorescent RT-PCR nucleic acids. Population Ⅲ is a placebo intramuscular injection of deltoid muscle of the upper arm.
  Interventions: Biological: Biological/Vaccine: Recombinant new coronavirus vaccine (CHO cells) placebo group

INTERVENTIONS:
Biological: Biological/Vaccine: Recombinant new coronavirus vaccine (CHO cell) low-dose group — Intramuscular injection of deltoid muscle of upper armof 25μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population I
Biological: Biological/Vaccine: Recombinant new coronavirus vaccine (CHO cells) high-dose group — Intramuscular injection of deltoid muscle of upper armof 50μg/0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population II
Biological: Biological/Vaccine: Recombinant new coronavirus vaccine (CHO cells) placebo group — Intramuscular injection of deltoid muscle of upper armof 0.5ml/person doseRecombinant new coronavirus vaccine (CHO cells).
  Arms: Population Ⅲ

SUMMARY:
Popular topic: Phase I clinical trial of recombinant new coronavirus vaccine (CHO cell) (≥60 years old) Research purpose: Main purpose: To evaluate the safety and tolerability of different doses of recombinant new coronavirus vaccine (CHO cells) in healthy people aged 60 years and above. Secondary purpose: to initially explore the immunogenicity and durability of different doses of recombinant new coronavirus vaccine (CHO cells).

Overall design: A single-center, randomized, double-blind, placebo-controlled trial design was adopted.

Study population: a healthy population of 60 years and above, a total of 50 cases, both men and women.

Test groups: 20 cases in the low-dose group, 5 cases in the placebo group; 20 cases in the high-dose group, 5 cases in the placebo group.

DETAILED DESCRIPTION:
Popular topic: Phase I clinical trial of recombinant new coronavirus vaccine (CHO cell) (≥60 years old) Product name: Recombinant new coronavirus vaccine (CHO cell),Each dose contains 25μg/0.5mL/bottle (low dose), 50μg/0.5mL/bottle (high dose) Indications: Prevention of respiratory diseases caused by new coronavirus infection Research population: healthy people ≥60 years old Research Unit: Hunan Provincial Center for Disease Control and Prevention Research purpose: Main purpose: To evaluate the safety and tolerability of different doses of recombinant new coronavirus vaccine (CHO cells) in healthy people aged 60 years and above. Secondary purpose: to initially explore the immunogenicity and durability of different doses of recombinant new coronavirus vaccine (CHO cells).

Overall design: A single-center, randomized, double-blind, placebo-controlled trial design was adopted.

Immunization program: 0, 1, and 2 months. Dose: Divided into low-dose group (25μg/0.5mL) and high-dose group (50μg/0.5mL).

Study population: a healthy population of 60 years and above, a total of 50 cases, both men and women.

Test groups: 20 cases in the low-dose group, 5 cases in the placebo group; 20 cases in the high-dose group, 5 cases in the placebo group.

Research plan and implementation:Volunteers aged 60 and above signed the informed consent form and asked about medical history, residence history and other information and then performed relevant examinations, including height, weight, vital signs, physical examination, laboratory tests (blood routine, urine routine, blood biochemistry), urine Pregnancy (women of childbearing age). After the study number is assigned, the subjects will collect throat swabs for SARS-CoV-2 real-time fluorescent RT-PCR nucleic acid detection, and blood will be collected for SARS-CoV-2 IgM and IgG antibody detection. Subjects will be in accordance with 0, 1, and 2 months Vaccination procedures are carried out. According to the order of the dose from low to high, it is divided into two stages and inoculated sequentially. Among them, placebo/five people per dose group, test vaccine/20 people per dose group, and qualified subjects were randomly enrolled into the test vaccine group and the placebo control group. In the first phase, subjects in the low-dose group (20 cases) and the placebo group (5 cases) were randomly enrolled; the safety data of the first 7-day vaccination was evaluated by DSMB, and if the suspension/termination criteria were not met, the first In the second-phase study, subjects in the high-dose group (20 cases) and the placebo group (5 cases) were randomly enrolled. Follow-up to 30 days after each dose, if the suspension/termination criteria is reached, DSMB will decide whether to inoculate the follow-up doses; in other cases, the investigator will decide whether to inoculate the follow-up doses.

Safety endpoint:

1. The incidence of all AEs within 1 month after the first dose to the full course of vaccination:

1. Total AE incidence;
2. The incidence of AEs related to research vaccines;
3. The incidence of grade 3 and above AE;
4. The incidence of grade 3 and above AEs related to research vaccines;
5. The incidence of AEs leading to withdrawal;
6. The incidence of AEs related to research vaccines leading to withdrawal; 2. The incidence of all serious adverse events (SAE) and the incidence of SAE related to the vaccine within 12 months after the first dose to the full course of vaccination; 3. Changes in the clinical significance of the laboratory test indicators after each dose of inoculation compared to before the first dose.

Immunogenicity endpoint:

Humoral immunity: before the first dose of vaccination, 1 month and 6 months after the full vaccination, neutralizing antibodies of novel coronavirus (SARS-CoV-2), S protein binding antibody (IgG), RBD protein binding antibody (IgG) ) Positive rate; The levels of neutralizing antibodies against SARS-CoV-2, S protein binding antibody (IgG) and RBD protein binding antibody (IgG) and their relative immunity 1 month and 6 months after the full vaccination of all subjects Increase the multiple before.

ELIGIBILITY:
standard constrain：

1. Persons with full capacity for civil conduct aged ≥60 years;
2. Subjects voluntarily agree to participate in the research and sign an informed consent form, and can provide valid identification; understand and comply with the requirements of the trial protocol; have the ability to understand (non-illiterate) research procedures and participate in the planned follow-up;
3. Axillary body temperature <37.3℃;
4. Female subjects and male subjects of childbearing age agree to take effective contraceptive measures during the study period.

Exclusion criteria：

1. The results of physical examination and laboratory examination before screening are abnormal and clinically significant as judged by clinicians, or systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg before screening;
2. A history of severe allergies to any component of the test vaccine, including aluminum preparations, such as: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis (Arthus reaction), dyspnea, blood vessels Neuroedema, etc.; or any previous history of serious side effects after the use of any vaccine or drug;
3. People with a history of SARS and SARS-CoV-2 (meet any of the following: ①Have a history of SARS and SARS-CoV-2 infection or onset; ②During this SRAS-CoV-2 epidemic, there are patients who have been diagnosed with the new crown/ Suspected patient contact history);
4. Have taken antipyretic or analgesic within 24 hours before the first dose of vaccination;
5. Inoculate subunit vaccine and/or inactivated vaccine within 14 days before the first dose of vaccine, and inoculate live attenuated vaccine within 30 days;
6. People suffering from the following diseases:

   * Acute (within 72 hours) feverish illness;

     * Suffering from digestive system diseases (such as diarrhea, abdominal pain, vomiting, etc.) in the past 7 days;

       * Suffering from congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;

         * Congenital or acquired immunodeficiency or autoimmune disease history or receiving immunomodulator treatment within 6 months, such as hormones; or monoclonal antibodies; or thymosin; or interferon, etc.; but local medication (such as ointment, Eye drops, inhalation or nasal spray);

           * Known to have been diagnosed with infectious diseases, such as: tuberculosis, viral hepatitis and/or human immunodeficiency virus HIV antibody positive or syphilis specific antibody positive;

             * Neurological diseases or neurodevelopmental dysfunction (for example, migraine, epilepsy, stroke, seizures in the last three years, encephalopathy, focal neurological deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis; History of mental illness or family history;

               ⑦Functional asplenia, as well as any cause of aspleen or splenectomy;

               ⑧Severe chronic diseases or conditions that cannot be controlled smoothly in the advanced stage, such as diabetes and thyroid disease;

               ⑨Severe liver and kidney diseases; respiratory diseases that currently require daily drug treatment (for example, chronic obstructive pulmonary disease [COPD], asthma) or any treatment for exacerbation of respiratory diseases (for example, asthma exacerbation) in the last 5 years; suffering from severe History of cardiovascular disease (such as congestive heart failure, cardiomyopathy, ischemic heart disease, arrhythmia, conduction block, myocardial infarction, pulmonary heart disease) or myocarditis or pericarditis;

               ⑩Have thrombocytopenia, any coagulation dysfunction or receive anticoagulant treatment, etc.;

               ?Tumor patients;
7. Have received blood or blood-related products, including immunoglobulin, within 3 months; or plan to use it during the research period;
8. Those who are already pregnant (including a positive urine pregnancy test), or are breastfeeding;
9. Any research or unregistered products (drugs, vaccines, biological products or devices) other than research products have been used within 3 months, or planned to be used during the research period;
10. The investigator believes that any disease or condition in the subject may put the subject at an unacceptable risk; the subject cannot meet the requirements of the protocol; it interferes with the assessment of the vaccine response.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of adverse events after intramuscular injection | 12 months after full vaccination
  The main observation methods of adverse reactions mainly include laboratory examination, local reactions and systemic reactions at the administration site.
Immunogenic end point | Within 6 months after the last dose of vaccination
  The positive rate of neutralizing antibody, S protein binding antibody (IgG), RBD protein binding antibody (IgG) of all subjects before the first dose, 1 month and 6 months after the full vaccination And titer levels and their fold increase before immunity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Xiangtan, Changsha, China

IPD SHARING:
Plan to Share IPD: No